CLINICAL TRIAL: NCT05465720
Title: "Invisible" Balance Problems: the Comparison of Effects of Motor, Sensory and Cognitive Exercises on Falls Prevention in Community Dwelling Older Adults
Brief Title: Comparison of Effects of Motor, Sensory and Cognitive Exercises on Falls Prevention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Huiya Chen, associate professor, Chung Shan Medical University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2022-07-17; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Motor, Sensory, Cognition, Older, Falls, Balance Ability, Randomized Controlled Trial, Task-oriented Approach

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- motor (Active Comparator)
  Interventions: Behavioral: falls-prevention programs
- sensory (Experimental)
  Interventions: Behavioral: falls-prevention programs
- cognitive (Experimental)
  Interventions: Behavioral: falls-prevention programs

INTERVENTIONS:
Behavioral: falls-prevention programs — Each group will receive 10-minute warm up, followed by 20-minute exercises in the ICF body function level, 20-minute exercises in the ICF activity level, and finally 10-minute cool down. The 10-minute war up include dynamic mobility exercises of the upper extremity and trunk (ribbons dancing on a chair) and of the lower extremity (marching in place). The 10-minute cool down include flexibility exercises of multiple muscles especially focusing on neck, hamstring, and calf muscles.

SUMMARY:
Motor, sensory, and cognitive functions all contribute to balance maintenance, and age causes deterioration in these functions with associated declines in balance ability and accidental falls. Relatively speaking, the sensory and cognitive functions are "invisible" in designing falls-prevention programs. The relative proportions of training of motor, sensory, and cognitive functions, for the most efficient falls-prevention program is a practical and important issue but has not been studied yet by directly comparing their intervention effects.

This three-year project aims to provide evidence base for relative proportions of motor, sensory, and cognitive training when designing falls-prevention programs. The crossover randomized controlled trial (RCT) will recruit 120 community-dwelling elderly adults from local community centers. There will two experimental groups- sensory and cognitive training, one control group- motor training, each for 60 minutes per session, 3 times a week, for 16 weeks. The three groups will be trained with task-oriented design of balance exercise but focusing on different aspects, i.e., training will begin in the ICF body function level (focusing on motor, sensory, or cognitive function) in the stance position and will end in the ICF activity level (balance or mobility activities focusing on motor, sensory, or cognitive function). The primary outcome measures are rates of falls and near-falls in the ICF participation level, and the secondary measures are balance/mobility performance and risk of falling in the ICF activity level.

In Taiwan, a great amount of expense is paid to prevent falls in the community setting. Through better understanding of the comparative intervention effects between motor, sensory, and cognitive training, this project hope to be able to suggest the relative proportions of motor, sensory, and cognitive training in falls-prevention exercise design.

ELIGIBILITY:
Inclusion Criteria:

* (1) older than 60 years of age, (2) living in the community, (3) scored more than two in Mini-Cog assessment [51], and (4) able to walk independently or with minimal assistance in the community

Exclusion Criteria:

* (1) an injury or musculoskeletal system disorder that would hamper their ability to conduct the physical tests, (2) acute heart attack in recent 3-6 months or unstable angina, (3) uncontrolled atrial or ventricular arrhythmias, (4) aortic dissecting aneurysm, (5) severe aortic stenosis, (6) acute endocarditis/pericarditis, (7) uncontrolled blood pressure higher than 180/110 mmHg, (8) acute thromboembolism, (9) acute or severe heart failure, (10) acute or severe respiratory failure, (11) uncontrolled postural hypotension, (12) uncontrolled acute decompensated diabetes mellitus or low blood sugar, (13) any other circumstance the doctors believe prevents dosing physical activity.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Short form of Falls Efficacy Scale International | 5 minutes
  Participants will be asked to report their concerns about falling from 1 to 4 when performing seven activities, including indoor activities, outdoor activities, and social events
Taiwan International Physical Activity Questionnaire-Short Form | 10 minutes
  The frail criterion of the minimum weekly energy expenditure is 383 Kcal for men and 270 Kcal for women
Rate of falls | 3 minutes
  participants will be interviewed for their falls history in the previous year
Rate of near-falls | 3 minutes
  participants will be interviewed for their falls history in the previous year